CLINICAL TRIAL: NCT07106593
Title: Treatment of TBI-Related Tinnitus and Comorbid PTSD: Examination of Neurobiological Markers Related to Symptom Improvement
Brief Title: Treatment for PTSD and Tinnitus
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00001126; HT9425-24-1-0988 (Other Grant/Funding Number: DoD CDMRP Traumatic Brain Injury and Psychological Health Research Program 2023)
Record Dates: First submitted 2025-06-27; First posted 2025-08-06 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: PTSD - Post Traumatic Stress Disorder; Posttraumatic Stress Disorder (PTSD); Tinnitus
Keywords: imaging; veterans; active duty; ptsd; tinnitus; treatment; cognitive processing therapy; cognitive behavioral therapy for tinnitus; military; psychotherapy; therapy; counseling
MeSH Terms: conditions — Combat Disorders; Stress Disorders, Post-Traumatic; Tinnitus

STUDY DESIGN:
Intervention Model Description: Participants will either receive Cognitive Processing Therapy (CPT) for PTSD first followed by Cognitive Behavioral Therapy for Tinnitus (CBT-t) for tinnitus; or vice versa: Cognitive Behavioral Therapy for Tinnitus (CBT-t) for tinnitus first followed by Cognitive Processing Therapy (CPT) for PTSD.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CPT-CBTt (Active Comparator): Participants will receive Cognitive Processing Therapy for PTSD followed by Cognitive Behavioral Therapy for Tinnitus
  Interventions: Behavioral: Cognitive Processing Therapy; Behavioral: CBT-t
- CBTt-CPT (Active Comparator): Participants will receive Cognitive Behavioral Therapy for Tinnitus followed by Cognitive Processing Therapy for PTSD
  Interventions: Behavioral: Cognitive Processing Therapy; Behavioral: CBT-t

INTERVENTIONS:
Behavioral: Cognitive Processing Therapy — CPT (Resick, Monson, & Chard, 2024) consists of 12 50-minute sessions conducted over a 6- to 12-week period (Resick, Monson, & Chard, 2008). The three phases of CPT include psychoeducation, processing, and challenging beliefs and assumptions related to the trauma, oneself, and the world.
Behavioral: CBT-t — The standard CBT-t protocol is gathered from the Progressive Tinnitus Management (PTM) program, and includes psychoeducation about how tinnitus can develop. CBT-t includes using behavioral principles to help manage tinnitus reactions, including the use of sounds: soothing sounds, background sound, and interesting sound. CBT-t teaches relaxation exercises, scheduling pleasant activities, and learn how to modify thoughts related to tinnitus. Therapists will also provide basic education on how to protect hearing health among participants in order to prevent worsening of tinnitus and to prevent exacerbation of any hearing loss.

SUMMARY:
In this study, researchers are examining the best sequence of interventions for posttraumatic stress disorder (PTSD) and tinnitus. Participants will either receive psychotherapy for PTSD first (Cognitive Processing Therapy; CPT), followed by treatment for tinnitus (Cognitive Behavioral Therapy for Tinnitus; CBT-t); or vice-versa. We also aim to identify changes in brain functioning after receiving therapy.

DETAILED DESCRIPTION:
After consenting to this study, study participants will be asked to speak with a study staff member about stressful or traumatic experiences, complete hearing assessments and questionnaires about exposure to traumatic events, PTSD symptoms, mental and physical health problems, such as depression and substance use, head injuries, and tinnitus. Participants who are able and willing may be asked to provide functional magnetic resonance imaging (MRI) scans before and after treatment. Participants will receive treatment for tinnitus and posttraumatic stress disorder (PTSD) in one of two ways: Cognitive Processing Therapy (CPT) first and then Cognitive Behavioral Therapy for Tinnitus (CBT-t) OR CBT-t first, followed by CPT.

ELIGIBILITY:
Inclusion Criteria:

* Adult male and female active duty military personnel and veterans seeking treatment for PTSD
* Diagnosis of PTSD
* Person has experienced at least one mild traumatic brain injury (concussion)
* Ability to speak and read English
* Stable on any psychotropic medications
* Meets criteria for chronic subjective and bothersome tinnitus
* Chronic tinnitus is at least possibly related to head injury

Exclusion Criteria:

* Currently receiving other talk therapies
* Severe hearing loss that would prevent the participant from benefiting from therapy
* Current severe suicidal ideation
* Psychiatric hospitalization in the last 12 months
* Moderate to severe substance use that would prevent the participant form benefiting from therapy
* Current manic episode or psychotic symptoms requiring immediate stabilization or hospitalization
* Significant cognitive impairment
* Moderate to severe brain damage
* Neurobiological disorders
* Temporomandibular joint disorders and/or Meniere's disease that cause acute pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-08-08 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
PTSD Checklist | Baseline to 6-Month Follow-Up (approximately12 months)
  Assessment of PTSD Symptoms
Tinnitus Functional Index | Baseline to 6-Month Follow-Up (approximately12 months)
  Assessment of Tinnitus-Related Distress

CONTACTS AND LOCATIONS:
Overall Officials: John Moring, PhD, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- The University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
At the conclusion of this study, participants who signed the consent to have their data placed in the STRONG STAR Repository will be maintained under the UTHSCSA IRB-approved Repository protocol. For participants who decline participation in the STRONG STAR Repository, at the conclusion of the study their data will be de-identified and the data maintained in the Repository without identifiers. The IRB approved STRONG STAR Repository is a large comprehensive database of information, biological specimens and neuroimages related to the identification, assessment, and treatment of posttraumatic stress disorder (PTSD), insomnia, pain, and related behavioral health conditions. No biospecimen data is being collected in this study.
Supporting Information: Study Protocol, SAP
Time Frame: Unending: Beginning immediately after publication with no end date.